CLINICAL TRIAL: NCT02973581
Title: Influence of Surgical Pleth Index-guided Analgesia Using Different Techniques on the Perioperative Outcomes in Patients Undergoing Vitreoretinal Surgery Under General Anaesthesia: Randomised, Controlled Trial
Brief Title: SPI-directed Analgesia for Vitreoretinal Surgeries
Acronym: SPIVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Michał Stasiowski, Principal Investigator, Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SilesianMUKOAiIT2
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-07

CONDITIONS: Vitreoretinal Surgeries; Postoperative Nausea and Vomiting; Postoperative Pain
Keywords: Surgical Pleth Index (SPI); General Anaesthesia (GA),; Numerical Rating Scale (NRS); Adequacy of Anaesthesia (AoA); Peribulbar Block (PBB); Topical Analgesia (TA); Oculocardiac reflex (OCR); Postoperative nausea nad vomiting (PONV); paracetamol; metamizol
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dipyrone; Acetaminophen; Lidocaine; proxymetacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- metamizol (Experimental): analgesic drug
  Interventions: Drug: Metamizol; Drug: 0,5 % bupivacaine with of 2% lidocaine
- acetaminophen (Experimental): analgesic drug
  Interventions: Drug: Metamizol; Drug: 0,5 % bupivacaine with of 2% lidocaine; Drug: Proxymetacaine
- 0,5 % bupivacaine with of 2% lidocaine (Experimental): a volume of 5 ml of analgesic solution for regional peribulbar block
  Interventions: Drug: Acetaminophen; Drug: 0,5 % bupivacaine with of 2% lidocaine; Drug: Proxymetacaine
- Proxymetacaine (Experimental): topical analgesia
  Interventions: Drug: Acetaminophen; Drug: Proxymetacaine
- control group (Placebo Comparator): patients will receive no pre-emptive analgesia. standard doses of fentanyl will be used intraoperatively.
  Interventions: Drug: Metamizol; Drug: Acetaminophen; Drug: 0,5 % bupivacaine with of 2% lidocaine; Drug: Proxymetacaine

INTERVENTIONS:
Drug: Metamizol — in group A patients will receive pre-emptive analgesia using intravenous infusion of metamizol in a single dose of 1-1,25 gram
  Arms: acetaminophen; control group; metamizol
Drug: Acetaminophen — in group P patients will receive pre-emptive analgesia using intravenous infusion of acetaminophen in a single dose of 10-15 mg per kg of body weight
  Other Names: paracetamol
  Arms: 0,5 % bupivacaine with of 2% lidocaine; Proxymetacaine; control group
Drug: 0,5 % bupivacaine with of 2% lidocaine — in group PBB patients in group BF will receive regional peribulbar block using a solution of 0,5% bupivacaine (2,5 ml) with 2% lidocaine (2,5 ml)
  Other Names: Lidocaine
  Arms: 0,5 % bupivacaine with of 2% lidocaine; acetaminophen; control group; metamizol
Drug: Proxymetacaine — in group T patients will receive topical analgesia using a solution of 0,5% Alcaine
  Other Names: Alcaine
  Arms: 0,5 % bupivacaine with of 2% lidocaine; Proxymetacaine; acetaminophen; control group

SUMMARY:
The aim of this randomized trial is to assess the efficacy of SPI-directed analgesia for vitreoretinal surgeries (VRS), presence of PONV and oculocardiac reflex (OCR) and compare Numerical Rating Scale (NRS) with Surgical Pleth Index (SPI) for monitoring pain perception postoperatively.

Patients received general anaesthesia alone or combined with either preemptive analgesia using topical solution of 0,5% proxymetacaine or peribulbar block (0,5% bupivacaine with 2% lidokaine) or preemptive intravenous infusion of 1,0 g of metamizol or preemptive intravenous infusion of acetaminophen in a doseof 10-15mg/kg of body weight.

DETAILED DESCRIPTION:
Monitoring depth of anaesthesia using spectral entropy (SE) and quality of neuromuscular block are routine in modern anaesthesia, whereas monitoring of analgesia still requires further studies. Recently, the Surgical Pleth Index (SPI) was added as a surrogate variable showing the nociception-antinociception balance into abovementioned parametres constituting a novel approach in monitoring patients intraoperatively, known as adequacy of anaesthesia (AoA) or tailor-made anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study
* written consent to undergo general anaesthesia alone or combined with different techniques of pre-emptive analgesia and vitreoretinal surgery

Exclusion Criteria

* history of allergy to local anaesthetics or metamizole
* necessity of administration of vasoactive drugs influencing SPI monitoring
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
pain perception intraoperatively | intraoperatively
  The investigators will compare the efficacy of analgesia intraoperatively according to technique of analgesia used preoperatively. The investigators will administer a rescue dose of fentanyl intravenously in a dose of 1 mcg per kg of body weight in the case when SPI value increases over 15 points in SPI scale every 5 minutes until SPI value decreases back to baseline value. Additionally, the investigators will analyse rescue fentanyl consumption in abovementioned groups
oculocardiac reflex rate | intraoperatively
  The investigators will compare the rate of presence of OCR intraoperatively in studied groups

SECONDARY OUTCOMES:
pain perception postoperatively | up to one hour after discharge to postoperative unit.
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: either local peribulbar block or topical analgesia or intravenous infusion of either metamizol or acetaminophen. The investigators use NRS and compare it with SPI values.
PONV | up to one hour
  The investigators will compare the presence of PONV after emergence from GA in studied groups. The investigators will observe patients postoperatively and record any incidence of nausea or vomiting and in the abovementioned case the investigators will administer a standard dose of antiemetic drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
article in European Journal of Anaesthesiology in 2018, case reports

REFERENCES:
- [Background] Mandelcorn M, Taback N, Mandelcorn E, Ananthanarayan C. Risk factors for pain and nausea following retinal and vitreous surgery under conscious sedation. Can J Ophthalmol. 1999 Aug;34(5):281-5. PMID 10486687
- [Result] Gruenewald M, Herz J, Schoenherr T, Thee C, Steinfath M, Bein B. Measurement of the nociceptive balance by Analgesia Nociception Index and Surgical Pleth Index during sevoflurane-remifentanil anesthesia. Minerva Anestesiol. 2015 May;81(5):480-9. Epub 2014 Jul 17. PMID 25032676
- [Result] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Result] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Result] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604
- [Result] Jaichandran VV, Raman R, Gella L, Sharma T. Local anesthetic agents for vitreoretinal surgery: no advantage to mixing solutions. Ophthalmology. 2015 May;122(5):1030-3. doi: 10.1016/j.ophtha.2014.11.026. Epub 2015 Jan 10. PMID 25582785
- [Result] Ghali AM. The efficacy of 0.75% levobupivacaine versus 0.75% ropivacaine for peribulbar anesthesia in vitreoretinal surgery. Saudi J Anaesth. 2012 Jan;6(1):22-6. doi: 10.4103/1658-354X.93050. PMID 22412772
- [Result] Bahcecioglu H, Unal M, Artunay O, Rasier R, Sarici A. Posterior vitrectomy under topical anesthesia. Can J Ophthalmol. 2007 Apr;42(2):272-7. PMID 17392852
- [Result] Seidenari P, Santin G, Milani P, David A. Peribulbar and retrobulbar combined anesthesia for vitreoretinal surgery using ropivacaine. Eur J Ophthalmol. 2006 Mar-Apr;16(2):295-9. doi: 10.1177/112067210601600216. PMID 16703549
- [Result] Eberhart LH, Morin AM, Hoerle S, Wulf H, Geldner G. Droperidol and dolasetron alone or in combination for prevention of postoperative nausea and vomiting after vitrectomy. Ophthalmology. 2004 Aug;111(8):1569-75. doi: 10.1016/j.ophtha.2004.01.031. PMID 15288990
- [Result] Subramaniam R, Subbarayudu S, Rewari V, Singh RP, Madan R. Usefulness of pre-emptive peribulbar block in pediatric vitreoretinal surgery: a prospective study. Reg Anesth Pain Med. 2003 Jan-Feb;28(1):43-7. doi: 10.1053/rapm.2003.50032. PMID 12567343
- [Result] Fekrat S, Elsing SH, Raja SC, Campochiaro PA, de Juan E Jr, Haller JA. Eye pain after vitreoretinal surgery: a prospective study of 185 patients. Retina. 2001;21(6):627-32. doi: 10.1097/00006982-200112000-00010. PMID 11756886
- [Result] Calenda E, Olle P, Muraine M, Brasseur G. Peribulbar anesthesia and sub-Tenon injection for vitreoretinal surgery: 300 cases. Acta Ophthalmol Scand. 2000 Apr;78(2):196-9. doi: 10.1034/j.1600-0420.2000.078002196.x. PMID 10794256
- [Result] Sajedi P, Nejad MS, Montazeri K, Baloochestani E. Comparing the preventive effect of 2 percent topical lidocaine and intravenous atropine on oculocardiac reflex in ophthalmological surgeries under general anesthesia. Int J Prev Med. 2013 Nov;4(11):1258-65. PMID 24404359
- [Result] Calenda E, Quintyn JC, Brasseur G. Peribulbar anaesthesia using a combination of lidocaine, bupivocaine and clonidine in vitreoretinal surgery. Indian J Ophthalmol. 2002 Sep;50(3):205-8. PMID 12355695
- [Result] Page MA, Fraunfelder FW. Safety, efficacy, and patient acceptability of lidocaine hydrochloride ophthalmic gel as a topical ocular anesthetic for use in ophthalmic procedures. Clin Ophthalmol. 2009;3:601-9. doi: 10.2147/opth.s4935. Epub 2009 Nov 2. PMID 19898665